CLINICAL TRIAL: NCT06528730
Title: A Novel Surgical Criteria for Degenerative Cervical Myelopathy in Chinese Ethnicity
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Law Ka Pui Karlen, Principle Investigator, The University of Hong Kong
Other Study IDs: UW 23-242
Record Dates: First submitted 2024-07-07; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Degenerative Cervical Spinal Stenosis
Keywords: Degenerative cervical myelopathy; diagnosis; physical performance tests; surgeical criteria; functional deficits
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: DCM — Confirm degenerative cervical myelopathy by Orthopaedic surgeon and MRI

SUMMARY:
Degenerative Cervical Myelopathy (DCM) is an age-related irreversible degenerative disease predominantly affecting the elderly aged 50 and over. DCM is usually triggered by ossification of the posterior longitudinal ligament or ossification of ligamentum flavum or prolapsed intervertebral disc over the cervical spine. Specific clinical signs characterized the presence of cervical spinal cord compression; including Hoffmann's sign, Finger Escape Sign, Scapulohumeral Reflex, and Reverse Supinator Reflex. Hand numbness, clumsiness, and gait disturbance. These are featured clinical manifestations and well-known indicators for detailed clinical and radiographic investigation, such as Magnetic Resonance Imaging (MRI) for diagnosis and surgical planning.

Surgical intervention is considered to be the most effective treatment for DCM worldwide. It is the only evidence-based treatment to halt disease progression and allow modest improvement in function and quality of life. DCM progression is not specific to predict the timing for surgery, though it is still debated. Length of symptoms, pre-operative Modified Japanese Orthopaedic Association Scoring System for Cervical Myelopathy (mJOA) and physical performance are suggested as recovery predictors in DCM.

In current practice, the offer of surgical treatment is entirely based on the combination of the evidence of cord compression in Magnetic Resonance Imaging (MRI) and mJOA. DCM who are at risk of critical neurological deficits have a reduced anteroposterior diameter of the spinal canal less than 9 mm or cross-sectional area of the spinal cord less than 40 sq. mm; mJOA less than 13 with evidence of functional deterioration will be offered with surgical intervention. MRI and mJOA are used as the golden standard for the indication of surgical intervention in the aspect of radiological deformities and self- perceived functional deficits. The concern on the clinical predictor, the physical performance, was overlooked and lacked a compromised criterion in the physical performance tests for surgical decisions. Therefore, this study aims to develop DCM-specific criteria from physical performance tests in predicting the surgical indication for DCM in the Chinese population.

DETAILED DESCRIPTION:
Degenerative Cervical Myelopathy (DCM) is a prevalent degenerative spinal disease that often goes unnoticed by general clinicians due to its non-specific and subtle signs and symptoms in its early stages. Delayed identification of DCM may lead to poor surgical outcomes or permanent disability, impacting the quality of life of affected individuals.

Incoordination in hand and gait movements are early signs of DCM that worsen with disease progression. Despite validated performance tests for DCM, there is currently no objective criterion for functional deficits in aiding clinical decision-making for surgery or diagnosis.

To meet the pressing global need for objective functional criteria, this study aims to develop surgical criteria specific to DCM. This will involve using physical performance tests, in addition to evaluating MRI findings of cord compression, clinical signs, and the modified Japanese Orthopedic Association (mJOA). By expediting the surgical decision-making process, we hope to improve recovery outcomes for individuals with DCM worldwide

ELIGIBILITY:
Inclusion Criteria:

* MRI confirmed Chinese DCM surgical candidates
* All gender
* Older than 45 years old
* Independent walkers
* No previous cervical spinal surgery
* Cognitively capable of following instructions.

Exclusion Criteria:

* Active diagnosis of tuberculosis spine
* Lumbar spinal diseases
* Extra-pyramidal
* Cerebral or cerebellar disorders
* Peripheral neuropathies
* Previous spinal operations
* Unable to walk independently with or without aids
* Non-communicable subjects and cognitively incapable of expressing their symptoms clearly

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patient with Degenerative Cervical Myelopathy will be recruited in DKCH
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
10-second Grip and Release test (GR) | 24 months
  Counting the no. of grip-release repetitions made in 10 seconds
10-second Stepping Test (SST) - no. of steps made in 10 seconds | 24 months
  Counting the no. of stepping repetitions made in 10 seconds
Foot Tapping Test (FTT) | 24 months
  Counting the no. of foot taps repetitions made in 10 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Karlen Ka-pui Law, M. Phil, Principal Investigator — The University of Hong Kong
Locations (1):
- The Duchess of Kent Children's Hospital at Sandy Bay, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
IPD sharing is not expected

REFERENCES:
- [Result] Fehlings MG, Tetreault LA, Riew KD, Middleton JW, Aarabi B, Arnold PM, Brodke DS, Burns AS, Carette S, Chen R, Chiba K, Dettori JR, Furlan JC, Harrop JS, Holly LT, Kalsi-Ryan S, Kotter M, Kwon BK, Martin AR, Milligan J, Nakashima H, Nagoshi N, Rhee J, Singh A, Skelly AC, Sodhi S, Wilson JR, Yee A, Wang JC. A Clinical Practice Guideline for the Management of Patients With Degenerative Cervical Myelopathy: Recommendations for Patients With Mild, Moderate, and Severe Disease and Nonmyelopathic Patients With Evidence of Cord Compression. Global Spine J. 2017 Sep;7(3 Suppl):70S-83S. doi: 10.1177/2192568217701914. Epub 2017 Sep 5. PMID 29164035
- [Result] Hilton B, Tempest-Mitchell J, Davies B, Kotter M. Assessment of degenerative cervical myelopathy differs between specialists and may influence time to diagnosis and clinical outcomes. PLoS One. 2018 Dec 17;13(12):e0207709. doi: 10.1371/journal.pone.0207709. eCollection 2018. PMID 30557368
- [Result] Tetreault L, Kopjar B, Nouri A, Arnold P, Barbagallo G, Bartels R, Qiang Z, Singh A, Zileli M, Vaccaro A, Fehlings MG. The modified Japanese Orthopaedic Association scale: establishing criteria for mild, moderate and severe impairment in patients with degenerative cervical myelopathy. Eur Spine J. 2017 Jan;26(1):78-84. doi: 10.1007/s00586-016-4660-8. Epub 2016 Jun 24. PMID 27342612
- [Result] Yukawa Y, Nakashima H, Ito K, Machino M, Kanbara S, Kato F. Quantifiable tests for cervical myelopathy; 10-s grip and release test and 10-s step test: standard values and aging variation from 1230 healthy volunteers. J Orthop Sci. 2013 Jul;18(4):509-13. doi: 10.1007/s00776-013-0381-6. Epub 2013 Apr 6. PMID 23564077
- [Result] Pribble BA, Black CD, Larson DJ, Larson RD. An evaluation of the reliability of the foot-tapping test in a healthy sample. Foot (Edinb). 2021 Sep;48:101851. doi: 10.1016/j.foot.2021.101851. Epub 2021 Jul 12. PMID 34385026
- [Result] Nakashima H, Yukawa Y, Ito K, Machino M, Kanbara S, Morita D, Imagama S, Hamajima N, Ishiguro N, Kato F. Validity of the 10-s step test: prospective study comparing it with the 10-s grip and release test and the 30-m walking test. Eur Spine J. 2011 Aug;20(8):1318-22. doi: 10.1007/s00586-011-1733-6. Epub 2011 Mar 6. PMID 21380747
- [Result] Kalsi-Ryan S, Singh A, Massicotte EM, Arnold PM, Brodke DS, Norvell DC, Hermsmeyer JT, Fehlings MG. Ancillary outcome measures for assessment of individuals with cervical spondylotic myelopathy. Spine (Phila Pa 1976). 2013 Oct 15;38(22 Suppl 1):S111-22. doi: 10.1097/BRS.0b013e3182a7f499. PMID 23963009
- [Result] Machino M, Ando K, Kobayashi K, Morozumi M, Tanaka S, Ito K, Kato F, Ishiguro N, Imagama S. Cut off value in each gender and decade of 10-s grip and release and 10-s step test: A comparative study between 454 patients with cervical spondylotic myelopathy and 818 healthy subjects. Clin Neurol Neurosurg. 2019 Sep;184:105414. doi: 10.1016/j.clineuro.2019.105414. Epub 2019 Jul 5. PMID 31306894
- [Result] Yukawa Y, Kato F, Ito K, Horie Y, Nakashima H, Masaaki M, Ito ZY, Wakao N. "Ten second step test" as a new quantifiable parameter of cervical myelopathy. Spine (Phila Pa 1976). 2009 Jan 1;34(1):82-6. doi: 10.1097/BRS.0b013e31818e2b19. PMID 19127165